CLINICAL TRIAL: NCT04164043
Title: Efficacy of a Recreation Therapy Community Based Wellness Recovery Program for Individuals With Parkinson's Disease
Brief Title: Efficacy of a Recreation Therapy Wellness Recovery Program for Individuals With Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision made on 8/16/2021 due to difficult enrollment because of limited access for enrollees during the pandemic and changes in staff
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00040793
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease
Keywords: Recreation Therapy; Community Based; Movement Disorder; Wellness Recovery Program
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Intervention Model Description: All participants will enter a 14 week baseline data collection period followed by a 12-week Wellness Recovery Program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recreational Therapy Wellness Recovery Program Group (Experimental): All participants will enter a baseline data collection period for two weeks. They will then participate in a 12-week community-based Recreational Therapy (RT) Wellness Recovery Program (WRP) for individuals with Parkinson's disease (WRP).
  Interventions: Behavioral: Wellness Recovery Program

INTERVENTIONS:
Behavioral: Wellness Recovery Program — 12-week community-based recreation therapy
  Other Names: WRP

SUMMARY:
The Recreation Therapy Wellness Recovery Program conducts group classes which provide repetitive training of foundational skills designed specifically for those with Parkinson's Disease. The course will encourage bigger and faster movements (adapted from the Parkinson Wellness Recovery, PWR!Moves ® program) and education on optimal function.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate a currently active community-based Recreational Therapy (RT) Wellness Recovery Program (WRP) for individuals with Parkinson's disease (PD) to determine the efficacy of the treatment intervention. Since PD is a progressive, degenerative neurological disease, it is critical that individuals with this diagnosis remain as active as possible to slow down the progression of the disease, improve balance and strength, and increase health-related quality of life. The overall goal of this project is to determine the efficacy of a neuroplasticity physical activity program in terms of improving balance, improving health-related quality of life, reducing stress, and increasing satisfaction in exercise including social connectedness of group exercise. There is evidence that the neuroplasticity model may be a more effective type of intervention than traditional exercise programs in improving symptoms of PD. The neuroplasticity approach requires repetition of complex tasks that are high intensity and present a novel challenge. This type of intervention has been shown to improve motor and cognitive behaviors which are critical areas of decline for those with PD. The WRP program uses a comprehensive neuroplasticity-principled program that integrates exercise and wellness. The PI, Julie Bradwell, LRT/CTRS is a Certified Instructor for Parkinson Wellness Recovery Power Moves. The RT Wellness Recovery program at Wake Forest Baptist Health is modeled on the Parkinson Wellness Recovery Power Moves. Components within the program include the Parkinson Power Moves and the exercise 4 Brain Change. This study will be a 14-week study with the first two weeks of collecting baseline data and immediately following with a 12-week intervention program to increase balance, health-related quality of life, and satisfaction in exercise in individuals with PD as well as reduce stress. Most research on RT interventions for this population are in traditional settings (inpatient or rehabilitation settings). When discharged from these settings, many individuals become less active, have few social interactions and lose the benefits of exercise and physical therapy they gained while in these programs once they are home. The WRP community-based program at Wake Forest Baptist Health has the potential to prevent secondary complications as well as slow down the progression of the disease for participants. If the outcomes of this project suggest this type of intervention will improve the functional skills, quality of life, and/or satisfaction in exercise for individuals with PD and reduce stress, it will provide the RT discipline with evidenced based practice intervention for this population

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects in this study will have a diagnosis of Parkinson's disease.
* Potential subjects in this study are able to tolerate a 60-minute exercise program; participants complete the Parkinson Power Moves Class Application which requires a release form and a physician's signature that identifies any limitations or precautions to be taken in the program.

Exclusion Criteria:

* Individuals who do not have a diagnosis of Parkinson's disease or those with PD who are not medically cleared to participate in the program will be excluded.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Sit to Stand Test | Baseline Measure 1 performed at day 1 after signing consent
  Measures functional muscle strength in the lower limbs. This test is reported in seconds.
Sit to Stand Test | Baseline Measure 2 performed at day 2 after signing consent
  Measures functional muscle strength in the lower limbs. This test is reported in seconds.
Sit to Stand Test | Week 4 post baseline period
  Measures functional muscle strength in the lower limbs. This test is reported in seconds.
Sit to Stand Test | Week 8 post baseline period
  Measures functional muscle strength in the lower limbs. This test is reported in seconds.
Sit to Stand Test | Week 12 post baseline period
  Measures functional muscle strength in the lower limbs. This test is reported in seconds.
Timed Floor Transfer Test | Baseline Measure 1 performed at day 1 after signing consent
  Measures vestibular balance and functional mobility to determine risk of falling. This test is reported in seconds.
Timed Floor Transfer Test | Baseline Measure 2 performed at day 2 after signing consent
  Measures vestibular balance and functional mobility to determine risk of falling. This test is reported in seconds.
Timed Floor Transfer Test | Week 4 post baseline period
  Measures vestibular balance and functional mobility to determine risk of falling. This test is reported in seconds.
Timed Floor Transfer Test | Week 8 post baseline period
  Measures vestibular balance and functional mobility to determine risk of falling. This test is reported in seconds.
Timed Floor Transfer Test | Week 12 post baseline period
  Measures vestibular balance and functional mobility to determine risk of falling. This test is reported in seconds.
Timed Up and Go (TUG) test | Baseline Measure 1 performed at day 1 after signing consent
  Test involves a series of transitional movements including sit to stand, walking, turning and sit to stand. The test is reported in seconds.
Timed Up and Go (TUG) test | Baseline Measure 2 performed at day 2 after signing consent
  Test involves a series of transitional movements including sit to stand, walking, turning and sit to stand. The test is reported in seconds.
Timed Up and Go (TUG) test | Week 4 post baseline period
  Test involves a series of transitional movements including sit to stand, walking, turning and sit to stand. The test is reported in seconds.
Timed Up and Go (TUG) test | Week 8 post baseline period
  Test involves a series of transitional movements including sit to stand, walking, turning and sit to stand. The test is reported in seconds.
Timed Up and Go (TUG) test | Week 12 post baseline period
  Test involves a series of transitional movements including sit to stand, walking, turning and sit to stand. The test is reported in seconds.
The Blue Foam (stand) with Trek Poles Test | Baseline Measure 1 performed at day 1 after signing consent
  Test involves lateral moves and front and back moves with or without assistance. measures level of assistance needed: supervision or modified assistance.
The Blue Foam (stand) with Trek Poles Test | Baseline Measure 2 performed at day 2 after signing consent
  Test involves lateral moves and front and back moves with or without assistance. measures level of assistance needed: supervision or modified assistance.
The Blue Foam (stand) with Trek Poles Test | Week 4 post baseline period
  Test involves lateral moves and front and back moves with or without assistance. measures level of assistance needed: supervision or modified assistance.
The Blue Foam (stand) with Trek Poles Test | Week 8 post baseline period
  Test involves lateral moves and front and back moves with or without assistance. measures level of assistance needed: supervision or modified assistance.
The Blue Foam (stand) with Trek Poles Test | Week 12 post baseline period
  Test involves lateral moves and front and back moves with or without assistance. measures level of assistance needed: supervision or modified assistance.
Parkinson's Disease Questionnaire Short Form (PDQ8) | Baseline Measure 1 performed at day 1 after signing consent
  This is a spcific health related quality of life instrument created for individuals with Parkinson's Disease. Likert scale (0 - 4), higher the score the greater the functioning. Overall score ranges from 0 -32. Higher scores indicate greater impact of the disease
Parkinson's Disease Questionnaire Short Form (PDQ8) | Baseline Measure 2 performed at day 2 after signing consent
  This is a spcific health related quality of life instrument created for individuals with Parkinson's Disease. Likert scale (0 - 4), higher the score the greater the functioning. Overall score ranges from 0 -32. Higher scores indicate greater impact of the disease
Parkinson's Disease Questionnaire Short Form (PDQ8) | Week 4 post baseline period
  This is a spcific health related quality of life instrument created for individuals with Parkinson's Disease. Likert scale (0 - 4), higher the score the greater the functioning. Overall score ranges from 0 -32. Higher scores indicate greater impact of the disease
Parkinson's Disease Questionnaire Short Form (PDQ8) | Week 8 post baseline period
  This is a spcific health related quality of life instrument created for individuals with Parkinson's Disease. Likert scale (0 - 4), higher the score the greater the functioning. Overall score ranges from 0 -32. Higher scores indicate greater impact of the disease
Parkinson's Disease Questionnaire Short Form (PDQ8) | Week 12 post baseline period
  This is a spcific health related quality of life instrument created for individuals with Parkinson's Disease. Likert scale (0 - 4), higher the score the greater the functioning. Overall score ranges from 0 -32. Higher scores indicate greater impact of the disease
Psychological Need Satisfaction in Exercise Scale (PNSES) | Baseline Measure 1 performed at day 1 after signing consent
  Total range 1-6. Lower scores denotes worse outcome.
Psychological Need Satisfaction in Exercise Scale (PNSES) | Baseline Measure 2 performed at day 2 after signing consent
  Total range 1-6. Lower scores denotes worse outcome.
Psychological Need Satisfaction in Exercise Scale (PNSES) | Week 4 post baseline period
  Total range 1-6. Lower scores denotes worse outcome.
Psychological Need Satisfaction in Exercise Scale (PNSES) | Week 8 post baseline period
  Total range 1-6. Lower scores denotes worse outcome.
Psychological Need Satisfaction in Exercise Scale (PNSES) | Week 12 post baseline period
  Total range 1-6. Lower scores denotes worse outcome.
Perceived Stress Scale (PSS-10) | Baseline Measure 1 performed at day 1 after signing consent
  Total range 0-4. Lower scores denotes worse/better outcome.
Perceived Stress Scale (PSS-10) | Baseline Measure 2 performed at day 2 after signing consent
  Total range 0-4. Lower scores denotes worse/better outcome.
Perceived Stress Scale (PSS-10) | Week 4 post baseline period
  Total range 0-4. Lower scores denotes worse/better outcome.
Perceived Stress Scale (PSS-10) | Week 8 post baseline period
  Total range 0-4. Lower scores denotes worse/better outcome.
Perceived Stress Scale (PSS-10) | Week 12 post baseline period
  Total range 0-4. Lower scores denotes worse/better outcome.
Pain Rating Scale | completed week 3 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 4 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 5 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 6 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 7 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 8 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 9 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 10 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 11 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 12 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 13 after signing consent
  10 point rating scale, low score indicates less pain.
Pain Rating Scale | completed week 14 after signing consent
  10 point rating scale, low score indicates less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Cromer, LRT, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT04164043/ICF_000.pdf